CLINICAL TRIAL: NCT01236170
Title: Understanding Quality and Equity in Wheelchairs for Veterans
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: B7148-I
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Results first posted 2014-12-31 (Estimated); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injuries; Amputees
Keywords: Amputees; spinal cord injuries; quality of life; satisfaction; healthcare disparities; wheelchairs
MeSH Terms: conditions — Spinal Cord Injuries; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Veterans with spinal cord injury or amputated limbs who use a wheelchair as their primary source of mobility

SUMMARY:
The Department of Veterans Affairs (VA) provides wheelchairs to about 42,000 Veterans with SCI and more than 40,000 Veterans with amputated limbs (AL). Despite VA's efforts to remove financial and other barriers to the provision of wheelchairs to all Veterans who need them, preliminary evidence suggests that disparities exist in the quality of wheelchairs prescribed to racial minorities and low income Veterans with SCI or AL. The proposed project will provide important information to the VA about the quality and equity of wheelchairs provided to Veterans with SCI or AL, and it will identify the patient and provider factors associated with wheelchair provision. Because Veterans with SCI and AL are considered special disability populations, identifying and understanding these factors is a critical first step to developing interventions to increase the quality and equity of wheelchairs provided to all disabled Veterans.

DETAILED DESCRIPTION:
Wheelchairs enable Veterans to participate in home, employment, and social activities that might otherwise be inaccessible to them, thereby improving their quality of life (QOL). Despite VA's efforts to remove financial and other barriers to the provision of high quality wheelchairs to all Veterans, preliminary evidence suggests that disparities exist in the quality of wheelchairs prescribed to vulnerable (e.g., minority race/ethnicity, lower socioeconomic status) Veterans with Spinal Cord Injury (SCI) or amputated limbs (AL). This finding is concerning because patients who receive lower quality wheelchairs may be at risk for adverse physical, psychological, economic, and QOL outcomes. Mounting research demonstrates that patient psychosocial characteristics (e.g., medical mistrust, perceived discrimination, locus of control) and provider factors (e.g., demographics and training) are associated with disparities in healthcare processes and outcomes. However, for Veterans with SCI or AL, no studies to date have examined (a) what patient and provider factors are associated with the prescription of high quality wheelchairs, and (b) how these factors are associated with wheelchair quality and patient outcomes. The proposed cross-sectional, multi-site study of Veterans with SCI or AL who use a wheelchair as their primary source of mobility aims to determine whether: (1) patient demographic (e.g., race, SES) and psychosocial characteristics (e.g., medical mistrust, experience of discrimination) and provider factors (e.g., years of practice, certification, demographics) are associated with wheelchair quality; (2) wheelchair quality is associated with key patient outcomes, including satisfaction with medical care, QOL, amount of wheelchair activity, and participation in social and work-related activities; (3) patient and provider factors are independently associated with key patient outcomes including satisfaction with medical care, QOL, amount of wheelchair activity, and participation; and (4) the association of patient and provider factors with patient outcomes is explained by differences in wheelchair quality. Veterans with SCI or AL, who were prescribed their wheelchairs through the VA, will be recruited from the Philadelphia, PA, Cleveland, OH, Richmond, VA, and Bronx, NY VA Medical Centers to participate in an interview to assess their demographic characteristics, health information, psychosocial characteristics (including, experience of discrimination, perceived racism, medical mistrust, self-image, anxiety/depression, health beliefs, health literacy, and communication) and health-related outcomes (including wheelchair skills, satisfaction, QOL, participation). We will also assess amount of wheelchair activity using data logging devices, and determine wheelchair quality by its make and model. Data will also be collected from all health care providers involved in wheelchair provision for study participants.

Provider factors will include demographics (e.g., race/ethnicity, age, gender), and specialty (i.e., MD/OT/PT).

For Occupational and Physical Therapists, we will determine if they are certified by the Rehabilitation Engineering and Assistive Technology Society of North America. Years of practice since completion of medical training, number of chairs prescribed over the span of their career, what role each provider plays in the wheelchair provision process, as well as the number of continuing medical education (CME) credits and/or educational credit units (ECU) they have obtained in the past 3 years related specifically to wheelchairs, will also be assessed. Understanding the associations among the proposed patient characteristics and provider factors is an essential step toward developing tailored interventions, aimed at patients and providers, to improve the quality and equity of wheelchair service delivery for Veterans.

ELIGIBILITY:
Inclusion Criteria:

Veterans

* age >18 years
* must have SCI with discernible neurological impairments or an amputated lower limb which results in the use of a wheelchair
* must be in power or manual wheelchair >1 year and treated at the participating VAMC
* participants must use a manual or power wheelchair as their primary means of mobility (e.g., use wheelchair > 40 hours/week
* and be non-ambulatory except for exercise purposes

Exclusion Criteria:

* In wheelchair less than 1 year
* Able to ambulate without the use of a wheelchair
* Other disorders requiring the use of a wheelchair (e.g., MS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the following four VA Medical Centers: the Philadelphia VA Medical Center in Philadelphia, PA; the Louis Stokes VA Medical Center in Cleveland, OH; The Hunter Holmes McGuire VA Medical Center in Richmond, VA; and the James J. Peters VA Medical Center in Bronx, NY. Recruitment will occur at SCI clinics, amputee clinics, wheelchair clinics, and patient registries.
Sampling Method: Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Myaskovsky, PhD, Principal Investigator — Center for Health Equity Research and Promotion
Locations (5):
- United States (5):
  - James A. Haley Veterans' Hospital, Tampa, FL, Tampa, Florida
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Center for Health Equity Research and Promotion, Pittsburgh, Pennsylvania
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia

REFERENCES:
- [Result] Hart-Hughes S, Highsmith MJ, Phillips SL, Groer S. A review of clinical outcome assessment instruments for gait, balance, and fall rish in persons with lower level extremity amputation. Topics in Geriatric Rehabilitation. 2014 Mar 31; 30(1):70-76.
- [Derived] Myaskovsky L, Gao S, Hausmann LRM, Bornemann KR, Burkitt KH, Switzer GE, Fine MJ, Phillips SL, Gater D, Spungen AM, Boninger ML. How Are Race, Cultural, and Psychosocial Factors Associated With Outcomes in Veterans With Spinal Cord Injury? Arch Phys Med Rehabil. 2017 Sep;98(9):1812-1820.e3. doi: 10.1016/j.apmr.2016.12.015. Epub 2017 Jan 25. PMID 28130083
- [Derived] Myaskovsky L, Gao S, Hausmann LRM, Bornemann KR, Burkitt KH, Switzer GE, Fine MJ, Phillips SL, Gater D, Spungen AM, Worobey L, Boninger ML. Quality and Equity in Wheelchairs Used by Veterans. Arch Phys Med Rehabil. 2017 Mar;98(3):442-449. doi: 10.1016/j.apmr.2016.09.116. Epub 2016 Oct 3. PMID 27713075

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 497
Completed | 482
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 482
Age, Customized [Number; unit: participants] — The sum of participants in all categories for this measure does not equal the overall number of baseline participants because 4 participants had missing data for this measure.
  participants
    <=18 years | 0
    Between 18 and 65 years | 327
    >=65 years | 151
Sex/Gender, Customized [Number; unit: participants] — The sum of participants in both categories for the measure does not equal to overall number of baseline participants because one participant had missing data for this measure.
  participants
    Female | 19
    Male | 462
Region of Enrollment [Number; unit: participants]
  United States | 482

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Assessed With the Veterans RAND 12 Item Health Survey (VR-12)
Description: The investigators will assess QOL with the Veterans RAND 12 Item Health Survey (VR-12) and two additional physical function items designed for patients with SCI. Eight QOL domains are assessed, including physical functioning, vitality, role limitations due to physical problems, role limitations due to emotional problems, bodily pain, general health, social functioning, and mental health. The VR-12 has been used extensively with Veterans in a variety of health domains and has shown to be reliable and valid in ambulatory care populations (Cronbach's alpha= .83-.85). The additional two items were added because previous research demonstrated that existing measures of physical function in the VR12 are not appropriate to patients with SCI and are not able to reveal differences in physical function among SCI patients. The investigators assessed physical QOL and mental QOL, both scales range from 0 (worst possible outcome) to 100 (best possible outcome).
Time Frame: Measured at baseline
Population: Only 468/482 participants were included in this analysis due to 14 participants having missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 468
units on a scale
  Physical Quality of Life Summary Score | 44.7 (7.7)
  Mental Quality of Life Summary Score | 43.6 (15.4)

2. Secondary Outcome: Satisfaction With Wheelchair Service Delivery
Description: The investigators assessed Satisfaction with Wheelchair Service Delivery using the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 is an 8-item, easily administered and scored measure of client satisfaction with services (e.g., "How would you rate the quality of service you have received?"). For the purpose of this study, the investigators asked patients to focus specifically on satisfaction with service at their SCI or AL wheelchair clinic. The scale is unidimensional, yielding a homogenous estimate of general satisfaction with services. It is scored by summing the individual items and produces a score ranging from 8-32, with higher scores indicating greater satisfaction. The CSQ-8 has been extensively used in a variety of healthcare settings, operates similarly across ethnic groups, and demonstrates excellent psychometric properties (Cronbach's alpha = .83-.93).
Time Frame: one time use, at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 482
units on a scale | 26.6 (5.5)

3. Secondary Outcome: Satisfaction With Prescribed Wheelchair
Description: We assessed Satisfaction with patients' prescribe wheelchair using the Quebec User Evaluation of Satisfaction with assistive Technology ( (QUEST). We used an 8-item subset of the QUEST to assess patients' satisfaction with their wheelchair. QUEST is the first and only standardized satisfaction assessment tool that was designed specifically for assistive technology devices. Its' development was based on major theoretical models of assistive technology. The QUEST has been widely cited and used in clinical and research settings, and demonstrates strong psychometric properties (Cronbach's alpha = .82). The 8 item subset focuses specifically on patients' satisfaction with different aspects of their wheelchair (e.g., "How satisfied are you with the dimensions (size, height, length, width) of your assistive device?"). Responses range from 1(not satisfied at all) to 5(very satisfied). Cronbach's alpha = .80 for the 8-item wheelchair subset. We chose to eliminate the other four items.
Time Frame: one time use, at baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 1
Number analyzed (Participants) | 482
units on a scale | 4.1 (0.9)

4. Secondary Outcome: Participation in Society
Description: We assessed participation in society with a modified version of the Craig Handicap Assessment and Reporting Technique Short Form (CHART-SF). The CHART was designed to provide a simple measure of involvement in life situations ("In a typical week, how many days do you get out of your house and go somewhere?") with sub-scales measuring physical independence, cognitive independence, mobility, occupation, social integration and economic self-sufficiency. The CHART-SF produces scores ranging from 0 (severe handicap) to 100 (no handicap) for each of the sub-scales and a total score ranging from 0-600. The CHART-SF is the most widely used participation measure in rehabilitation research. It has been used in various ethnic groups, and has well-established psychometric properties (test-retest reliability = .93; inter-rater reliability = .83). We dichotomized into "Disabled" and "Not Disabled" where disabled are those with a CHART score <100, and not disabled are those with a CHART score >=100
Time Frame: Measured at baseline
Population: 452/482 participants were included in this analysis because 30 participants had missing data.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 452
participants
  Disabled (<100) | 208
  Not Disabled (>=100) | 244

5. Secondary Outcome: Wheelchair Activity
Time Frame: over a two week period following baseline
Population: Access to data is no longer available.
Arm/Group | Group 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/497
Other Adverse Events (participants affected / at risk) | 0/497

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes